CLINICAL TRIAL: NCT04530136
Title: Recombinant Human C1 Esterase Inhibitor (Ruconest®) in the Prevention of Severe SARS-CoV-2 Infection in Hospitalized Patients With COVID-19: a Randomized, Parallel-group, Open-label, Multi-center Pilot Trial in the US
Brief Title: Prevention of Severe SARS-CoV-2 Infection in Hospitalized Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C1 6201
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Confirmed Coronavirus Disease
MeSH Terms: interventions — conestat alfa

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruconest (Experimental): Patients receive (150 U/ml) of Ruconest at a 50 U/kg dose (max dose of 4200 U) as a slow intravenous injection via a peripheral every 12 hours; for 4 days. A total of 8 doses will be administered.
  Interventions: Drug: Ruconest
- Standard of Care (Other): SOC
  Interventions: Drug: Ruconest

INTERVENTIONS:
Drug: Ruconest — Patients will be randomized to Ruconest or Standard of Care
  Other Names: SOC

SUMMARY:
The primary purpose of this study is to evaluate if adding rhC1-INH to standard of care (SOC) in patients admitted for stage II COVID-19 infection may reduce the risk of disease progression, i.e. ALI requiring mechanical ventilation, or increase the chance of a faster clinical improvement compared to SOC alone.

DETAILED DESCRIPTION:
Patients fulfilling all eligibility criteria will be randomized in a 2:1 ratio in an open-label controlled design to treatment with rhC1-INH in addition to SOC or SOC only starting on day 0. The first rhC1-INH treatment will be administered on the same day and continued for a total of 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years,
* Admitted to the hospital because of confirmed positive SARS-CoV-2 (COVID-19 infection).
* Evidence of pulmonary involvement on CT scan or X-Ray of the chest,
* Symptom onset within the previous 10 days AND at least one additional risk factor for progression to mechanical ventilation: 1) arterial hypertension, 2) >50 years, 3) obesity (BMI>30.0 kg/m2), 4) history of cardiovascular disease, 5) chronic pulmonary disease, 7) chronic renal disease, 6) C-reactive protein of >35mg/L, 7) oxygen saturation at rest in ambient air of <94%

Exclusion Criteria:

* Contraindications to the class of drugs under study (C1 esterase inhibitor);
* History or suspicion of allergy to rabbits;
* Women who are of childbearing potential and not using methods of contraception during the entire study period;
* Pregnant or breastfeeding females or has a positive serum β-human chorionic gonadotropin (hCG) pregnancy test at screening;
* Chronic liver disease (any Child-Pugh score B or C);
* Currently admitted to an ICU or expected admission within the next 24 hours; and
* Currently receiving invasive or non-invasive ventilation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bernstein, MD, Principal Investigator — University of Cincinnati
Locations (4):
- United States (4):
  - Virtua Marlton Hospital, Marlton, New Jersey
  - Virtua Memorial Hospital, Mount Holly, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Virtua Voorhees Hospital, Voorhees Township, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to two parallel groups in a 2:1 ratio to receive either rhC1INH (intervention) in addition to standard of care (SOC) or SOC treatment (control). Randomization was stratified by the study site before inclusion using randomly permuted block sizes of four.
Period: Overall Study
Arm/Group | Ruconest | Standard of Care
Started | 27 | 11
Completed | 24 | 7
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analyzed (FAS/ITT - Interim analysis/Overrunning analysis) in interim analysis phase: rhC1INH plus SOC [n=23]; SOC alone [n=9]. A subsequent (post hoc) analysis was conducted to include all 38 patients, overrunning analysis phase: rhC1INH plus SOC [n=27]; SOC alone [n=11].
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruconest | Standard of Care | Total
Number analyzed (Participants) | 27 | 11 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 7 | 30
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.93 (11.84) | 55.18 (8.99) | 55.55 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 16
  Male | 14 | 8 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 25 | 8 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.58 (6.07) | 30.54 (8.55) | 32.56 (7.31)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Each Score on WHO 7-point Outcome Scale at Day 7
Description: The disease severity on the 7-point WHO Ordinal Scale on Day 7 was the primary objective of this study. This endpoint had been suggested by the WHO for clinical trials in patients with Covid-19. The ordinal scale measures illness severity over time. The higher score, the worst outcome: meaning score 1, no limitation in activities and score 7, death.
Time Frame: Assessed on each day after enrollment (worst status) with the use of the WHO Ordinal Scale and the score on day 7 will be analyzed stratified by its baseline value
Measure: Count of Participants; unit: Participants
Arm/Group | Ruconest | Standard of Care
Number analyzed (Participants) | 27 | 11
Participants
  WHO ordinal scale 1 | 6 | 0
  WHO ordinal scale 2 | 20 | 8
  WHO ordinal scale 3 | 0 | 0
  WHO ordinal scale 4 | 1 | 0
  WHO ordinal scale 5 | 0 | 1
  WHO ordinal scale 6 | 0 | 2
Statistical Analysis 1: Comparison: Ruconest vs Standard of Care; Test type: Superiority; p = 0.0346, Wilcoxon rank test

2. Secondary Outcome: Time to Clinical Improvement
Description: Time from randomization to an improvement of (at least) two (score) points on the seven-category WHO Ordinal Scale or live discharge from hospital whichever came first within 14 days after enrollment
Time Frame: Daily until day 14
Measure: Mean (Standard Error); unit: days
Arm/Group | Ruconest | Standard of Care
Number analyzed (Participants) | 27 | 11
days | 3.32 (0.32) | 4.91 (1.43)
Statistical Analysis 1: Comparison: Ruconest vs Standard of Care; Test type: Superiority; p = 0.4441, WHO Ordinal Scale

3. Secondary Outcome: Invasive (Mechanical) or Non-invasive Ventilation
Description: Admission to ICU with invasive or non-invasive ventilation will be assessed.
Time Frame: Daily until day 14.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruconest | Standard of Care
Number analyzed (Participants) | 27 | 11
Participants
  Invasive (mechanical) ventilation | 0 | 2
  Non-invasive ventilation | 12 | 7
Statistical Analysis 1: Comparison: Ruconest vs Standard of Care; Test type: Superiority; p = 0.1021, WHO Ordinal Scale for Clin Improvement

4. Secondary Outcome: Number of Days Hospitalized
Description: Amount of days the patient is hospitalized during participation in the study.
Time Frame: between D0 and D90
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ruconest | Standard of Care
Number analyzed (Participants) | 27 | 11
days | 5.38 (1.76) | 11.27 (16.01)
Statistical Analysis 1: Comparison: Ruconest vs Standard of Care; Test type: Superiority; p = 0.1615, WHO Ordinal Scale

ADVERSE EVENTS:
Time Frame: From signing off ICF till 90 days follow-up period Adverse event date were collected.
Arm/Group | Ruconest | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/11
Serious Adverse Events (participants affected / at risk) | 3/27 | 2/11
Other Adverse Events (participants affected / at risk) | 23/27 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruconest (N=27) | Standard of Care (N=11)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood beta-D-glucan increased (Investigations) | 0 (0) | 1 (1)
Fibrin D Dimer increased (Investigations) | 1 (1) | 0 (0)
Transaminitis (Investigations) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure [Death] (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruconest (N=27) | Standard of Care (N=11)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase inc (Investigations) | 4 (4) | 1 (1)
C-reactive protein increased (Investigations) | 2 (2) | 1 (1)
Fibrin D dimer increased (Investigations) | 5 (5) | 1 (1)
Serum ferritin increased (Investigations) | 2 (2) | 1 (1)
Transaminitis (Investigations) | 6 (6) | 0 (0)
Interleukin level increased (Investigations) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT04530136/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT04530136/SAP_001.pdf